CLINICAL TRIAL: NCT00454038
Title: Preliminary Study of Hypro-Sorb® F Bilayer Bioabsorbable Membrane for Guided Tissue and Bone Regeneration
Brief Title: Study of Collagen Membrane in Guided Bone Regeneration
Acronym: GBR
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: watad sami, CARDIOPHIL LTD
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ae-01.CTIL
Record Dates: First submitted 2007-03-28; First posted 2007-03-29 (Estimated); Last update posted 2009-07-10 (Estimated); Status verified 2009-01

CONDITIONS: Cystectomy; Segmental Growing of Alveolar Tissue; Sinus Lift; Root Amputation and Apicoectomy; Periimplantitis
Keywords: cystectomy; augmentation; sinus; amputation; implant
MeSH Terms: conditions — Peri-Implantitis; Fistula

INTERVENTIONS:
Device: HYPRO SORB F — resorbable, double layered, collagen membrane

SUMMARY:
The main purpose of this study is to investigate the efficacy of Hypro-Sorb® F, a bilayered bioabsorbable membrane in inducing bone regeneration in different dental procedures requiring GBR.

DETAILED DESCRIPTION:
Guided bone regeneration is a procedure used in dentistry for the reconstruction of osseous defects around teeth, dental implants, and prior to implant placement. The main function of the membrane barrier in GBR is to mechanically prevent the undesirable penetration of epithelial cells and fibroblasts to the bone defect area, creating a secluded space where bone regeneration may occur. Resorbable and non-resorbable membranes have been used in GBR. While non resorbable membranes require another surgical procedure for removing the membrane after the healing period, the resorbable membranes have the advantage of transmitting tissue fluids, excluding undesirable cell penetration and sparing an additional unwanted surgical procedure. The aim of this study is to investigate the efficacy of Hypro-Sorb® F, a bilayered bioabsorbable membrane in inducing bone regeneration in different dental procedures requiring GBR.

ELIGIBILITY:
Inclusion Criteria:

* Cystectomy
* Segmental growing of alveolar tissue
* Lifting of the sinus bottom
* Root amputation
* Apicoectomy
* Filling of the alveolus after resections in prosthetic surgical practice
* Periimplantitis
* Maxillofacial surgery

Exclusion Criteria:

* Inside bone fractures when acrylate adhesives are applied.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-01 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
expected | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Alabuni Emad, Study Chair — The Baruch Padeh Medical Center
Locations (1):
- The Baruch Padeh Medical Center, Poriya, Tiberias, Israel